CLINICAL TRIAL: NCT00837785
Title: A 24-Hour Pharmacokinetic Determination of BG00012 After Single-Day Oral Administration in Subjects With Multiple Sclerosis
Brief Title: A 24-Hour Pharmacokinetic Determination of BG00012 After Single-Day Oral Administration in Subjects With MS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 109MS101
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Dimethyl Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 240 mg (two 120 mg capsules) twice a day
  Interventions: Drug: BG00012
- 2 (Experimental): 240 mg (two 120 mg capsules) three times a day
  Interventions: Drug: BG00012

INTERVENTIONS:
Drug: BG00012 — 240 mg (two 120 mg capsules) orally three times a day
  Arms: 2
Drug: BG00012 — 240 mg (two 120 mg capsules) orally twice a day
  Arms: 1

SUMMARY:
To establish a pharmacokinetic (PK) profile of BG00012, as measured by its primary metabolite, monomethyl fumarate (MMF), during a 24-hour dosing period in subjects with relapsing-remitting multiple sclerosis (RRMS), with a variety of baseline demographic characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 55 years old, inclusive, at the time of informed consent.
2. Have a confirmed diagnosis of RRMS according to McDonald criteria #1-4.
3. Be ambulatory.

Exclusion Criteria:

1. Primary progressive, secondary progressive, or progressive-relapsing multiple sclerosis (PRMS).
2. History of any clinically significant cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic (other than MS), dermatologic, psychiatric, renal, oncologic, anaphylaxis or other major diseases, as determined by the Investigator.
3. Current enrollment in any other drug, biologic, or device study or treatment with another investigational drug within 6 months or 5 half-lives of the investigational product, whichever time period is longer.
4. Serious infection (e.g., pneumonia, septicemia) within the 2 months prior to Day -1.
5. Pregnant or nursing women.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2009-02-28 (Actual); Primary Completion 2009-10-31 (Actual); Study Completion 2009-10-31 (Actual)

PRIMARY OUTCOMES:
To establish a PK profile of MMF during a 24-hour BG00012 dosing period in subjects with RRMS | 24 Hours

SECONDARY OUTCOMES:
To explore the relationship of differences in baseline demographics and dosing factors in the disposition of BG00012 | 24 Hours

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Berlin, Germany